CLINICAL TRIAL: NCT05195112
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of MT921 in Subjects With Moderate to Severe Submental Fat
Brief Title: Evaluate the Efficacy and Safety of MT921 in Subjects With Moderate to Severe Submental Fat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT11-KR19SMF309
Record Dates: First submitted 2021-12-13; First posted 2022-01-18 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Submental Fat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT921 (Experimental): * Injection volume/interval: 0.2mL/1.0cm
  * Number of Injection: Maximum 50 times
  * Concentration per unit area: 3mg/cm2
  Interventions: Drug: MT921
- Placebo (Placebo Comparator): * Injection volume/interval: 0.2mL/1.0cm
  * Number of Injection: Maximum 50 times
  * Concentration per unit area: 0mg/cm2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT921 — Active ingredient
  Arms: MT921
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of MT921 in Subjects with Moderate to Severe Submental fat compared with Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19~65 years of age
2. CA-SMFRS and PA-SMFRS score of 2 or 3
3. Satisfaction level is 3points or less
4. Voluntarily provide informed consent

Exclusion Criteria:

1. Following history that can affect the efficacy and safety evaluation in the chin or neck area as judged by the investigator

   * Scars or skin lesion on the study treatment region
   * Liposuction or lipolytic material treatment to decrease submental fat
   * Permanent filler, synthetic implantation and autologous fat grafting
   * Within 1 year of screening visit, semi-permanent filler (Calcium Hydroxyapatite, collagen-stimulator, etc.), radio-frequency treatment, HIFU, thread, laser procedure and chemical peeling procedure over medium-depth
   * Within 6 months of screening visit, temporary filler (Hyaluronic acid, etc.) procedure on the chin or neck, injection of botulinum toxin, radio-frequency treatment, HIFU, thread, laser procedure and chemical peeling procedure over medium-depth
2. BMI over 35.0 kg/m^2
3. Submandibular enlargement due to causes other than localized subcutaneous fat (hyperthyroidism, cervical lymphadenopathy, etc.)
4. Current or past dysphagia
5. Judged difficult to measure submandibular fat due to sagging skin on the chin and neck or wide platysmal bands on the neck
6. Bleeding or taking anticoagulant drugs (except for patients taking anticoagulant drugs, those who can discontinue administration from 3 days before injection to 24 hours after injection of the IP)
7. Skin disease or would infection on the study treatment region
8. Hypersensitivity to Lidocaine, Benzocaine, Procaine or the IP
9. Pregnancy or breast feeding or female of child-bearing potential who has not agreed to use of medically acceptable contraception during the study period

   * All women of childbearing age have negative pregnancy test results can be enrolled in parallel with surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or menopause (amenorrhea for more than 12 months).
   * Medically acceptable contraception: Intrauterine device, Intrauterine system, vasectomy, tubal ligation, condom, Cervical cap, Contraceptive diaphragm, contraceptive sponges, spermicide, oral contraceptive pill and etc.
10. Experience of other clinical trials within 30 days before screening
11. Any other clinically meaningful conditions that are considered ineligible for the study in the medical judgement of principal investigator or sub-investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose CA-SMFRS (Clinician-Assessed Submental Fat Rating Scale) score changed | 12 weeks
  Proportion of subjects whose CA-SMFRS decreased 1, 2 points or more compared the 12 weeks after the last administration day to before administration of the IP, Minimum value: 0 (best outcome) / Maximum value: 4 (worst outcome)
Proportion of subjects whose PA-SMFIS (Patient Assessed-Submental Fat Impact Scale) score changed | 12 weeks
  Proportion of subjects whose PA-MFRS decreased 1, 2 points or more compared the 12 weeks after the last administration day to before administration of the IP , Minimum value: 0 (worst outcome) / Maximum value: 10 (best outcome)

SECONDARY OUTCOMES:
Proportion of subjects whose CA-SMFRS (Clinician-Assessed Submental Fat Rating Scale) score changed | 4 weeks
  Proportion of subjects whose CA-SMFRS decreased 1, 2 points or more compared the 4 weeks after the last administration day to before administration of the IP, Minimum value: 0 (best outcome) / Maximum value: 4 (worst outcome)
Proportion of subjects whose PA-SMFIS (Patient Assessed-Submental Fat Impact Scale) score changed | 4 weeks
  Proportion of subjects whose PA-MFRS decreased 1, 2 points or more compared the 4 weeks after the last administration day to before administration of the IP , Minimum value: 0 (worst outcome) / Maximum value: 10 (best outcome)
PA-SMFIS (Patient Assessed-Submental Fat Impact Scale) | 4 and 12 weeks
  Change PA-SMFIS (Patient Assessed-Submental Fat Impact Scale) score compared 4 to 12 weeks after the last administration of the IP, Minimum value: 0 (worst outcome) / Maximum value: 10 (best outcome)
Measuring submental fat volume by MRI (magnetic resonance imaging) | 12 weeks
  Confirmation the volume of submental fat compared the 12 weeks after the last administration to before administration of the IP measured by MRI (Number of Participants: approximately 120)
Satisfaction Evaluation by the subject | 4 and 12 weeks
  A score of 5 (slightly satisfied) or higher in the subject satisfaction evaluation at 4 and 12 weeks after the last administration to before administration of the IP

OTHER OUTCOMES:
Caliper | 4 and 12 weeks
  Percentage of change in submental fat thickness as measured by Caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided